CLINICAL TRIAL: NCT03705936
Title: Inducing Metaplasticity in Human Pharyngeal Motor Cortex Through Preconditioned Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Metaplasticity in Human Pharyngeal Motor Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor of Neurogastroenterology, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-4900-7208
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Deglutition; Physiology
Keywords: Non-invasive brain stimulation; Swallowing; Metaplasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Sham 1Hz rTMS--5Hz rTMS (Sham Comparator): Participants will receive sham 1Hz rTMS, then immediately followed by 5Hz rTMS.
  Interventions: Device: rTMS
- 1Hz rTMS--5Hz rTMS (Experimental): Participants will receive 1Hz rTMS, then immediately followed by 5Hz rTMS.
  Interventions: Device: rTMS
- 1Hz rTMS--30-minute break--5Hz rTMS (Experimental): Participants will receive 1Hz rTMS, then followed by 30 minutes break, then followed by 5Hz rTMS.
  Interventions: Device: rTMS
- 1Hz rTMS--60-minute break--5Hz rTMS (Experimental): Participants will receive 1Hz rTMS, then followed by 60 minutes break, then followed by 5Hz rTMS.
  Interventions: Device: rTMS
- Sham 5Hz rTMS--1Hz rTMS (Sham Comparator): Participants will receive sham 5Hz rTMS, then immediately followed by 1Hz rTMS.
  Interventions: Device: rTMS
- 5Hz rTMS--1Hz rTMS (Experimental): Participants will receive 5Hz rTMS, then immediately followed by 1Hz rTMS.
  Interventions: Device: rTMS
- 5Hz rTMS--45-minute break--1Hz rTMS (Experimental): Participants will receive 5Hz rTMS, then followed by 45 minutes break, then followed by 1Hz rTMS.
  Interventions: Device: rTMS
- 5Hz rTMS--90-minute break--1Hz rTMS (Experimental): Participants will receive 5Hz rTMS, then followed by 90 minutes break, then followed by 1Hz rTMS.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — rTMS is a non-invasive brain stimulation technique. It can regulate brain activities with electrical pulses sent to the brain through electromagnetic induction.

SUMMARY:
The purpose of the study is to determine the effects of giving 2 doses of brain stimulation through repetitive transcranial magnetic stimulation (rTMS) on swallowing neurophysiology (brain function) in healthy adults.

DETAILED DESCRIPTION:
Recent studies have suggested that repetitive transcranial magnetic stimulation (rTMS), which is a well-established and tried and tested non-invasive (no surgical procedures involved) brain stimulation technique that can vary brain activities, may be used as a treatment for patients with swallowing difficulties. However, results have also showed that the response to the treatment is different among individuals. A possible explanation for this variation is related to the brain's level of activity preceding rTMS. The hypothesis of this study is that this variation may be minimized by regulating the brain state with an additional dose of rTMS prior to the intended rTMS session (preconditioned rTMS). This may subsequently improve the outcomes of rTMS.

Therefore, this study aims to better regulate the response of the brain to rTMS. The findings of this study will provide the basis for future development of optimal rTMS treatment protocols for patients with swallowing difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 years old or above; and
* No medical complications or significant past medical history

Exclusion Criteria:

* History of epilepsy;
* Previous history of neurosurgery;
* Previous swallowing problem;
* Implanted brain electrodes, cardiac pacemaker; or
* Use of medications (predominantly taking multiple anti-depressants) that lower neural threshold

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Pharyngeal motor evoked potentials (PMEPs) | Change from baseline up to 150 minutes after rTMS
  Motor evoked potentials from the pharynx will be elicited by single pulse transcranial magnetic stimulation and recorded.
Thenar (hand) motor evoked potentials (TMEPs) | Change from baseline up to 150 minutes after rTMS
  Motor evoked potentials from the hand will be elicited by single pulse transcranial magnetic stimulation and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, PhD, FRCP, Principal Investigator — The University of Manchester
Locations (1):
- Salford Royal Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No